CLINICAL TRIAL: NCT04540549
Title: Effects of Exercise on Patients With Functional Dyspepsia Based on Rome IV Criteria
Brief Title: Effects of Exercise on Functional Dyspepsia Based on Rome IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020031
Record Dates: First submitted 2020-08-29; First posted 2020-09-07 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Functional Dyspepsia
Keywords: functional dyspepsia, exercise, Rome IV
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Jogging or cycling ≥5 days/week, 30-60 min/d
  Interventions: Behavioral: exercise
- control group (No Intervention): The control group was encouraged to maintain their lifestyle.

INTERVENTIONS:
Behavioral: exercise — Jogging or cycling ≥5 days/week, 30-60 min/d
  Arms: intervention group

SUMMARY:
Functional dyspepsia is one of the most common gastrointestinal disorders (FGIDs) encountered in clinical practice. Functional dyspepsia is a clinical syndrome characterized by chronic and recurrent gastroduodenal symptoms in the absence of any organic or metabolic disease that is likely to explain the symptoms. Functional dyspepsia has a high incidence in the population. A recent research showed that FD is present in 11% of the Italian general population. It dramatically reduces a patient's quality of life, with an economic impact due to frequent clinical consultations, medication, and time off work. Although some experts recommend exercise as a first-line treatment for functional dyspepsia, there is little data on the relationship between exercise and functional dyspepsia, which needs to be confirmed by further research. Investigators designed this randomized controlled study to assess the effect of exercise on patients with functional dyspepsia based on Rome IV criteria.

DETAILED DESCRIPTION:
Functional dyspepsia is one of the most common gastrointestinal disorders (FGIDs) encountered in clinical practice. Functional dyspepsia is a clinical syndrome characterized by chronic and recurrent gastroduodenal symptoms in the absence of any organic or metabolic disease that is likely to explain the symptoms. Functional dyspepsia has a high incidence in the population. A recent research showed that FD is present in 11% of the Italian general population. It dramatically reduces a patient's quality of life, with an economic impact due to frequent clinical consultations, medication, and time off work.

Regular physical activity and exercise may be a way of life to reduce low levels of inflammation throughout the body, thereby reducing the risk of developing chronic diseases. Multiple studies have shown that after regular exercise, markers of inflammation and oxidative stress are reduced, while markers of inflammation and antioxidants are increased, reflecting the anti-inflammatory and antioxidant properties of exercise.

Rome IV was introduced in 2016. Rome IV introduced more precisely define the minimal thresholds for frequency and severity of each individual symptom, primarily for scientific purposes, but data still need to be collected to define thresholds based on the frequency and/or severity of symptoms that impair quality of life.

Although some experts recommend exercise as a first-line treatment for functional dyspepsia, there is little data on the relationship between exercise and functional dyspepsia, which needs to be confirmed by further research. Investigators designed this randomized controlled study to assess the effect of exercise on patients with functional dyspepsia based on Rome IV criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Functional dyspepsia meeting Rome IV criteria
3. Gastroscope, blood routine, liver function and Hp examination were performed within the last year, and the results were normal
4. No prokinetic drug, proton pump inhibitor or mucosal protective agent was used in the last two weeks
5. Sign informed consent and be willing to participate in this study

Exclusion Criteria:

1. There are organic diseases that may explain the symptoms, such as peptic ulcer, gastrointestinal neoplasms, history of hepatobiliary and pancreatic diseases, history of tumor diseases, and history of metabolic diseases
2. Pregnancy, prepregnancy, or lactation
3. History of abdominal surgery
4. Mental illness
5. Severe impairment of heart, liver, or kidney function or respiratory function
6. Recent use of antidepressant, hormone, NSAIDs
7. The main symptoms are gastroesophageal reflux disease or irritable bowel syndrome
8. Failure to increase exercise levels

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Weekly global symptom assessment | 12 weeks
  Patients are asked to answer the following yes/no question once a week: "In the past 7 days, have you had adequate relief of your stomach symptoms?"

SECONDARY OUTCOMES:
Eight items of dyspepsia symptom score questionnaire(epigastric pain, epigastric burning, postprandial fullness, early satiety, belching, bloating, nausea, and vomiting) | 12 weeks
  severity(0=absent; 1=mild; 2=moderate); frequency (1 = less than once per week; 2 = once per week; 3 = two to three times per week; 4 = four to five times per week; 5 = daily)
  3=severe and interfering with daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Wang, MD, Study Director — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China

IPD SHARING:
Plan to Share IPD: No